CLINICAL TRIAL: NCT02145195
Title: Food-based Solutions for Optimal Vitamin D Nutrition and Health Through the Life Cycle (ODIN) Junior
Brief Title: The Effect of Vitamin D Supplements on Vitamin D Status, Cardiometabolic Health and Immune Defense in Danish Children
Acronym: ODIN Junior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University College Cork (Other); University of Surrey (Other)
Responsible Party: Principal Investigator, Christian Mølgaard, MD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D214; European Commission (Other Grant/Funding Number: Contract no. 613977)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Children; Supplements; Cardiometabolic markers; Immune defense; Bone turnover; Muscle strength
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D (10 microgram/day) (Experimental): Tablets with 10 microgram vitamin D3 (cholecalciferol) daily for 20 weeks.
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Vitamin D (20 microgram/day) (Experimental): Tablets with 20 microgram vitamin D3 (cholecalciferol) daily for 20 weeks.
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Placebo control (Placebo Comparator): Tablets with 0 microgram vitamin D daily for 20 weeks.

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol)
  Arms: Vitamin D (10 microgram/day); Vitamin D (20 microgram/day)

SUMMARY:
The main purpose of this study is to investigate whether and in which doses vitamin D intake is needed in order to maintain an adequate vitamin D status in 4-8 year-old Danish children during wintertime.

DETAILED DESCRIPTION:
The main objective of ODIN Junior is to investigate whether and in which doses vitamin D intake is needed in order to maintain serum 25(OH)D concentrations above deficiency and insufficiency cut-offs (30 nmol/L and 50 nmol/L, respectively) in 4-8 year-old Danish children during the winter time. The children will be randomized to receive tablets with either 10 micrograms/day or 20 microgram/day of vitamin D3 (cholecalciferol), corresponding to one and two times the recommended daily intake in children, or placebo for 20 weeks. Measurements and blood sampling will be performed before the beginning and by the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 4-8 years at the start of the intervention
* healthy
* of white, Danish/European origin
* children must be Danish-speaking
* parents must read and speak Danish
* not planning a winter vacation south of a latitude of 51°North (corresponding to Surrey, England)

Exclusion Criteria:

* diseases that may interfere with vitamin D or calcium metabolism
* intake of medication known to affect vitamin D or calcium metabolism
* use of vitamin D containing supplements ≥ 4 days/week the last 8 weeks before intervention start and use of any vitamin D containing supplements the last 4 weeks before intervention start
* concomitant participation in other studies involving dietary supplements or blood sampling
* serum calcium > 2.7 mmol/L at baseline

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D status | Baseline and 20 weeks
  Serum concentrations of total 25-hydroxyvitamin D [25(OH)D]

SECONDARY OUTCOMES:
Change in anthropometric measurements | Baseline and 20 weeks
  Waist circumference, body weight, height, body mass index (BMI) and BMI z-scores.
Change in body composition | Baseline and 20 weeks
  Fat mass, fat mass index (kg/m2), fat free mass and fat free mass index (kg/m2).
Serum calcium | Baseline and 20 weeks
  Serum calcium (adjusted for albumin) evaluated after the first visit has been completed for all children, and after the second visit.

OTHER OUTCOMES:
Change in cardio-metabolic markers | Baseline and 20 weeks
  Blood pressure, insulin, cholesterols etc.
Change in markers of immune defense | Baseline and 20 weeks
  Production of cytokines in whole blood cultures. Expression of immune markers and antiviral and antimicrobial peptides.
Change in muscle strength | Baseline and 20 weeks
  Maximum hand grip strength.
Dietary intake of vitamin D and calcium | Baseline and 20 weeks
  Assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mølgaard, PhD, MD, Principal Investigator — Section of Peadiatric and International Nutrition, Department of Nutrition, Exercise and Sports, University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Mortensen C, Molgaard C, Hauger H, Kristensen M, Damsgaard CT. Sun behaviour and physical activity associated with autumn vitamin D status in 4-8-year-old Danish children. Public Health Nutr. 2018 Dec;21(17):3158-3167. doi: 10.1017/S1368980018002094. Epub 2018 Sep 7. PMID 30189911
- [Derived] Hauger H, Molgaard C, Mortensen C, Ritz C, Frokiaer H, Smith TJ, Hart K, Lanham-New SA, Damsgaard CT. Winter Cholecalciferol Supplementation at 55 degrees N Has No Effect on Markers of Cardiometabolic Risk in Healthy Children Aged 4-8 Years. J Nutr. 2018 Aug 1;148(8):1261-1268. doi: 10.1093/jn/nxy080. PMID 29917069
- [Derived] Mortensen C, Molgaard C, Hauger H, Kristensen M, Damsgaard CT. Winter vitamin D3 supplementation does not increase muscle strength, but modulates the IGF-axis in young children. Eur J Nutr. 2019 Apr;58(3):1183-1192. doi: 10.1007/s00394-018-1637-x. Epub 2018 Feb 15. PMID 29450728
- [Derived] Mortensen C, Damsgaard CT, Hauger H, Ritz C, Lanham-New SA, Smith TJ, Hennessy A, Dowling K, Cashman KD, Kiely M, Molgaard C. Estimation of the dietary requirement for vitamin D in white children aged 4-8 y: a randomized, controlled, dose-response trial. Am J Clin Nutr. 2016 Nov;104(5):1310-1317. doi: 10.3945/ajcn.116.136697. Epub 2016 Oct 12. PMID 27733403